CLINICAL TRIAL: NCT07192406
Title: Cross-cultural Adaptation of the Toxic Masculinity Scale Among Nursing Students in Indonesia: A Psychometric Testing Study
Brief Title: Cross-cultural Adaptation of the Toxic Masculinity Scale Among Indonesian Nursing Students: A Psychometric Testing
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Yudisa Diaz Lutfi Sandi, Principal Investigator, Kaohsiung Medical University
Other Study IDs: 25.7.24
Record Dates: First submitted 2025-07-24; First posted 2025-09-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Masculinity; Nursing; Scale Reliability Validity; Student
Keywords: nursing; masculinity; student; psychometry; scale
MeSH Terms: conditions — Masculinity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to adapt and validate the Toxic Masculinity Scale (TMS) for use among nursing students in Indonesia, ensuring its cultural relevance and psychometric soundness. The process involved cross-cultural adaptation through translation, expert review, and pilot testing, followed by psychometric evaluation using a sample of Indonesian nursing students.

DETAILED DESCRIPTION:
This study aimed to adapt and validate the Toxic Masculinity Scale (TMS) for use among nursing students in Indonesia, ensuring its cultural relevance and psychometric soundness. The process involved cross-cultural adaptation through translation, expert review, and pilot testing, followed by psychometric evaluation using a sample of Indonesian nursing students.

Key steps included: Translation and back-translation of the original scale, Content validation by experts in gender studies and nursing education, Exploratory and confirmatory factor analyses (EFA & CFA) to test construct validity and Reliability testing using Cronbach's alpha for internal consistency

ELIGIBILITY:
Inclusion Criteria:

* nursing student
* more than 17 years
* fluent in the Indonesian language

Exclusion Criteria:

* catastropic condition
* gap year during study

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all nursing students are in indonesia national wide
Sampling Method: Non-Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2025-09-23 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Toxic Masculinity | one time
  The Toxic Masculinity Scale (TMS-28) measures endorsement of harmful masculine norms across four domains: Masculine Superiority, Gender Rigidity, Emotional Restriction, and Repressed Suffering. Higher scores indicate stronger beliefs in male dominance, rigid gender binaries, emotional suppression, and avoidance of help when in pain. In validation samples, average scores were around 58 (on a 28-140 range), suggesting generally low-to-moderate endorsement. The scale demonstrated excellent reliability (α ≈ .93) and strong validity, correlating positively with traditional masculinity norms and negatively with feminist attitudes. These outcomes help identify patterns of toxic masculinity that may impact well-being and relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Novi S Nursafitri, RN, Principal Investigator — School of Health Science, Politeknik Negeri Subang
Locations (1):
- School of Health Science, Politeknik Negeri Subang, Subang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will not be shared due to confidentiality concerns and ethical restrictions outlined in the informed consent process. Participants were assured that their data would only be used for the purposes of this study and would not be shared publicly or with third parties.

REFERENCES:
- [Result] Sanders SM, Garcia-Aguilera C, Borgogna NC, Sy JRT, Comoglio G, Schultz OAM, Goldman J. The Toxic Masculinity Scale: Development and Initial Validation. Behav Sci (Basel). 2024 Nov 14;14(11):1096. doi: 10.3390/bs14111096. PMID 39594396
- [Result] Parent MC, Gobble TD, Rochlen A. Social Media Behavior, Toxic Masculinity, and Depression. Psychol Men Masc. 2019 Jul;20(3):277-287. doi: 10.1037/men0000156. Epub 2018 Apr 23. PMID 38250140
- [Result] Jbilou J, Levesque N, Sonier RP, Tully PJ, Pinette-Drapeau I, Sonier V, Charbonneau A, Greenman PS, Grenier J, Chomienne MH. Canadian French Translation and Preliminary Validation of the Conformity to Masculine Norms Inventory: A Pilot Study. Am J Mens Health. 2021 Nov-Dec;15(6):15579883211057391. doi: 10.1177/15579883211057391. PMID 34836484
- [Result] Levant RF, McDermott R, Parent MC, Alshabani N, Mahalik JR, Hammer JH. Development and evaluation of a new short form of the Conformity to Masculine Norms Inventory (CMNI-30). J Couns Psychol. 2020 Oct;67(5):622-636. doi: 10.1037/cou0000414. Epub 2020 Feb 3. PMID 32011153